CLINICAL TRIAL: NCT03367845
Title: Efficacy of Family Programs for Improving Child and Family Health and Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Julia Braungart-Rieker, Professor and Head, Colorado State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: NotreDame; R01HD087319 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2017-12-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Behavior, Infant
Keywords: Parent sensitivity; Fathers; Attachment; Marital communication
MeSH Terms: conditions — Infant Behavior | interventions — Sensitivity and Specificity

STUDY DESIGN:
Intervention Model Description: 2 X 2 factorial design testing two different interventions
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care Providers and Assessors represent two different teams of staff. Each is blind to the other status (how families did during assessment and which group families are assigned to). They do not have access to each others' files.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Experimental): Phone contacts with content not focusing on sensitivity or couples' relationships
  Interventions: Behavioral: Control
- Sensitivity Intervention (Experimental): Home visits to enhance mother-infant and father-infant parental sensitivity; with COVID-19, we now conduct remote visits using Zoom
  Interventions: Behavioral: Sensitivity Intervention
- Couples Intervention (Experimental): Home visits to enhance constructive couples' communication; with COVID-19, we now conduct remote visits using Zoom
  Interventions: Behavioral: Couples' Intervention
- Sensitivity and Couples Intervention (Experimental): Home visits combining sensitivity and couples' interventions; with COVID-19, we now conduct remote visits using Zoom
  Interventions: Behavioral: Sensitivity and Couples' Intervention

INTERVENTIONS:
Behavioral: Control — Parents receive 8 phone contacts (1 per week) that do not focus on material in the sensitivity and couples communication intervention.
  Arms: Control
Behavioral: Sensitivity Intervention — 4 home visits take place. Mothers and fathers are video recorded with their infant (separately) for approximate 10-15 minutes at the beginning of each visit. The recorded situations are natural (e.g., playing together, bathing the baby, mealtime, etc.) and the family coach (interventionist) is not actively involved in the parent-child interaction. A different theme is covered across the four intervention sessions. For each parent-infant interaction recording, the family coach reviews the recordings between visits and provides feedback to parents in the following intervention session. The exception to this is that video of parent-child interactions during the lab pre-test is used for material at the first home visit. Each session takes approximately 90 minutes. Visits occur over an 8 week period with phone contacts between each session. Because of COVID-19, we now conduct remote visits using Zoom.
  Other Names: Videofeedback to Promote Positive Parenting
  Arms: Sensitivity Intervention
Behavioral: Couples' Intervention — The psycho-educational inter-parental conflict prevention curriculum is a 4-session program that takes place in the families' homes. Each session lasts approximately 90 minutes and involves discussion and practice of four themes pertinent to improving conflict process, communication, and emotional security in the family: Conflict Overview, Interparental Conflict and Children, Stresses of Parenting, and Emotional Security. The family coach scaffolds and supports the couples' development of constructive conflict behaviors. Visits occur over an 8 week period with phone contacts between each session. Because of COVID-19, we now conduct remote visits using Zoom.
  Arms: Couples Intervention
Behavioral: Sensitivity and Couples' Intervention — This group receives both the Sensitivity and Couples' Intervention in their home. There are 8 home visits (4 for Sensitivity and 4 for Couples Intervention). Because of COVID-19, we now conduct remote visits using Zoom.
  Arms: Sensitivity and Couples Intervention

SUMMARY:
The proposed research is relevant to public health because of the critical importance of infant attachment and early experiences to the lifetime trajectory of mental health and socio-emotional functioning. This Randomized Clinical Trial addresses major gaps in available family-wide programs that can promote healthy development that best serve infants, mothers, fathers, and inter-parental relationships in cost-effective ways. This study also systematically tests for which families the interventions are most effective and rigorously tests the theoretical processes that link changes in mother-infant, father-infant, and mother-father interactions with infant and parent outcomes.

DETAILED DESCRIPTION:
Preventative interventions involving video-feedback programs to promote parenting (VIPP) have been shown to be successful in improving maternal sensitivity and infant-mother attachment security. However, interventions might be substantially more effective if broader elements of family systems were also addressed, including father-child and inter-parental relationships, particularly given the growing body of evidence that highlights the importance of father involvement and positive engagement in children's socio-emotional development. Infancy is a particularly sensitive and vulnerable period not only for the child but also for the parents who often experience heightened daily stress, parenting demands, work-family role strain, and inter-parental discord associated with changes in the family.The proposed longitudinal study addresses major gaps by testing the effectiveness of family-wide preventative interventions designed to promote healthy development and functioning in infants, mothers, and fathers, including low-income families. This three-phase study involves a rigorous randomized clinical trial (RCT) approach and will involve a demographically diverse sample of 400 families. Phase I involves a lab and home pre-test (infants 6 months of age) and 8-week intervention period; Phase II (12 months) includes an initial post-test, and Phase III (16-18 months) involves a second post-test. Families will be randomly assigned to one of four conditions: sensitivity intervention (SI), couples intervention (CI), both (SI + CI) or control. Specific aims of the study include: (1) An evaluation of the effectiveness of the SI, CI, and SI+CI interventions at improving parental sensitivity, parental efficacy, parenting stress, inter-parental conflict, infant affective development, attachment security, behavior problems, and socio-emotional competence; (2) A test of the mechanisms through which change in behavior occurs. For example, relations between SI participation in Phase I and child attachment in Phase III may be mediated by enhanced parent sensitivity in Phase II.

Relations between CI participation and child outcomes may be mediated by inter-parental functioning and more effective communication skills; (3) An examination of factors that moderate the effectiveness of the interventions, determining which families benefit the most. Potential moderators include demographic characteristics, family (dis)organization, parents' own caregiving history, parents' depressive and anxious systems, and infant negative temperament; (4) Mother-father comparisons on direct effects, mediating mechanisms and moderating processes. This study builds upon past research towards increasing children's emotional security in multiple family relationships by testing new directions in preventative interventions in infancy, addressing the mother-child, father-child, and mother-father relationships. The goal is to foster children's socio-emotional development and security through cost-effective family-wide interventions in infancy that promote sensitive parent-infant interactions and improved inter-parental communication.

ELIGIBILITY:
Inclusion Criteria:

* Parents cohabiting
* Both mothers and fathers agree to participate
* Healthy infants with no known health problems

Exclusion Criteria:

* Discovery of developmental delays or health problems in infants

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parental Sensitivity | 12-months
  Observational measure of parent sensitivity during infant-parent interactions
Change in Child Care Activities Scale | 12-months
  Parent-report questionnaire assessing degree of involvement with infants at home, reflecting percent time engaging in each activity. Subscales include: Direct Care, Indirect Care, Play Activities, and Total score all ranging from 0 - 100. Higher values mean higher percentage of time spent in that caretaking activity. Scores are averaged to create the subscales and total score.
Change in Parenting Stress Index - Short Form Version III | 12 months
  Parent-report questionnaire assessing degree of stress about roles as a parent. Subscales include: Parental Distress (scale range from 5 - 60; 33 and higher = 85th percentile); Parent-Child Dysfunctional Interaction (scale range 5 - 60; 26 and higher = 85th percentile); Difficult Child (scale range 5 - 60; 33 and higher = 85th percentile); Total Score (scale range 15 - 180; 86 and higher = 85th percentile). Higher values mean greater levels of parenting stress. Scores are summed to create subscales and the total score.
Change in Parenting Sense of Competence Scale | 12-months
  Parent-report measure of self-efficacy in their role as a parent. Subscales include Satisfaction (cale range 9 - 54); Efficacy (scale range 8 - 48). Total Score (scale range 17 - 102). Higher values indicate a greater satisfaction, efficacy, and total sense of competence. Scores are summed to create the subscales and total score.
Change in Spousal Attachment Questionnaire | 12-months
  Parent report questionnaire assessing parents' security in their relationships with each other. Subscales include Preoccupied Attachment (scale range 1 - 7); Fearful Attachment (scale range 1 - 7); Secure Attachment (scale range 1 - 7). Higher values mean greater levels of that type of attachment to spouse. Scores are averages of item sets.
Change in Conflict and Problem Solving Scale | 12-months
  Parent report questionnaire assessing conflict strategies in spousal relationship. Subscales include Cooperation (scale range 0 - 36); Avoidance and Capitulation (scale range 0 - 60); Stonewalling (scale range 0 - 42); Verbal Aggression (scale range 0 - 48); Physical Aggression (scale range 0 - 42); Child Involvement (scale range 0 - 30); Conflict Resolution (scale range 0 - 39). Higher scores indicate greater levels of use of conflict strategies or greater resolution. Item sets are summed to create subscale scores.
Change in O'Leary Porter Scale | 12-months
  Parent report questionnaire assessing children's exposure to marital conflict. There is a total score (scale range 0 - 36). Higher values indicate more conflict. Items are summed to create the total score.
Change in Brief Infant Toddler Emotional Assessment | 12-months
  Parent questionnaire evaluating children's behavior problems and competence. Subscales include Problems (scale range 0 - 66); Competencies (scale range 0 - 22); Externalizing problems (scale range 0 - 12); Internalizing (scale range 0 - 16); Dysregulation (scale range 0 - 16); Autism Spectrum Disorder (scale range 0 - 17). Higher scores indicate higher levels of each construct or higher screening value for Autism Spectrum Disorder. Scores are summed.
Mother-Infant Attachment | 12 months
  Observational ratings of infant attachment security with mothers from the Strange Situation; with COVID-19, we no longer do in-person assessments so we now use a modified version of the Attachment Q-Sort which is an interview with mothers over zoom.
Father-Infant Attachment | 10 months
  Observational ratings of infant attachment security with fathers from the Strange Situation; with COVID-19, we no longer do in-person assessments so we now use a modified version of the Attachment Q-Sort which is an interview with fathers over zoom.
Change in Couples' communication styles | 12-months
  Observational measure of parents' conflict styles during discussions
Change in Infant Affect Regulation | 12-months
  Observational measure of infants' affective and regulatory behaviors during parent-child interactions and during couples' discussions

CONTACTS AND LOCATIONS:
Overall Officials: Julia Braungart-Rieker, Ph.D., Principal Investigator — Colorado State University; E M Cummings, Ph.D., Principal Investigator — University of Notre Dame
Locations (2):
- United States (2):
  - Fort Wayne Center for Children and Families, Fort Wayne, Indiana
  - William J. Shaw Center for Children and Families, South Bend, Indiana

IPD SHARING:
Plan to Share IPD: No
At the close of the study, subject data will be deidentified and individual participant data will no longer be available for further use.